CLINICAL TRIAL: NCT02285491
Title: Efficacy of Local Anesthetic Injection Into Both Angles of the Rectus Sheath Incision for Postoperative Cesarean Delivery Analgesia.
Brief Title: Local Anesthetic Injection Into Both Angles of the Rectus Sheath Incision
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, dr mohammed elsafty, Dr Mohammed Elsafty, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: els7680
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Cesarean Delivery Pain
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- bupivacaine group (Experimental): This is the group of patients that will receive 10ml of bupivacaine 0.5% injection in both angles of the rectus sheath incision
  Interventions: Drug: 10ml of bupivacaine 0.5%
- saline group (Placebo Comparator): This group will receive saline injections as placebo into both angles of the rectus sheath incision
  Interventions: Drug: Placebo
- bupivacaine and saline group (Experimental): This group will receive saline injection in one angle and 10ml of bupivacaine 0.5% injection in the opposite angle.
  Interventions: Drug: 10ml of bupivacaine 0.5%; Drug: Placebo

INTERVENTIONS:
Drug: 10ml of bupivacaine 0.5% — This is a local anesthetic that will be used to block the ilioinguinal nerve to alleviate pain at the wound site after lscs
  Arms: bupivacaine and saline group; bupivacaine group
Drug: Placebo — 10 ml of saline will be injected as a placebo and the investigator and the patient and the data assessor are all blinded to what the patients received.
  Other Names: saline
  Arms: bupivacaine and saline group; saline group

SUMMARY:
Local anesthetic will be injected into both angles of the rectus sheath incision in an attempt to block sensory nerves in this area that cause the sensation of pain from lscs wound.

ELIGIBILITY:
Inclusion Criteria:

* patients booked for lscs
* primisection
* singleton pregnancy

Exclusion Criteria:

* emergency cesarean section
* bleeding tendency
* hypersensitivity to local anesthetic

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain assessment during rest and ambulation by visual analogue scale | for 24 hours after lscs

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt